CLINICAL TRIAL: NCT07393295
Title: Evaluation of the Efficacy and Tolerability of a Transcutaneous Electrical Nerve Stimulation (TENS) Device for the Management of Endometriosis-associated Pain
Brief Title: Efficacy and Tolerability of TENS in Endometriosis-related Pain
Acronym: ELECTRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monath Electronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-A02028-41; AU 2080 (Other: CPP (Comité de protection des personnes Sud-Est VI))
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Pain Associated With Endometriosis or Adenomyosis; Pelvic Pain Associated With Refractory Endometriosis; Endometriosis
MeSH Terms: conditions — Adenomyosis; Endometriosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional TENS Group (Experimental): Conventional TENS for 4 weeks
  Interventions: Device: Conventional TENS
- Microstimulation TENS (Active Comparator): Microstimulation TENS for 4 weeks
  Interventions: Device: Microstimulation TENS

INTERVENTIONS:
Device: Conventional TENS — Every TENS treatment lasts for 45 minutes
  Arms: Conventional TENS Group
Device: Microstimulation TENS — Every TENS treatment lasts for 45 minutes
  Arms: Microstimulation TENS

SUMMARY:
ELECTRE is a single-center, randomized, prospective, longitudinal, controlled, two-arm, single-blind study lasting 4 weeks (P1 investigation phase) after a 4-week run-in period.

The study is followed by a 4-week extension phase (P2) in which all participants will be treated with active TENS.

Randomization will be balanced according to a 1:1 ratio.

DETAILED DESCRIPTION:
* Endometriosis is defined by the presence of endometrial tissue outside the uterine cavity. It affects 6% to 10% of women of childbearing age. Depending on its location, a distinction is made between superficial endometriosis, adenomyosis, and deep endometriosis. The potential mechanisms of endometriosis are still under discussion.
* Endometriosis is accompanied by a painful triad combining dysmenorrhea, dyspareunia, and chronic pelvic pain.
* Pain requires treatment due to its multiple impacts in terms of quality of life, anxiety, depression, loss of productivity at work, and absenteeism.
* Approximately one-third of women with endometriosis continue to suffer despite medical treatment.
* The pain of endometriosis is multifactorial, involving inflammatory, nociceptive, neuropathic, neurovascular, myofascial, and hormonal mechanisms. The recurrence of endometriosis-related pain means that it must be considered a chronic pain syndrome leading to peripheral and central neural sensitization. The intensity of the pain is not correlated with the severity of the disease.
* Transcutaneous electrical nerve stimulation (TENS) is a non-invasive, easy-to-use, well-tolerated, self-administered technique widely used for its analgesic effect in acute and chronic pain. Several studies have suggested the effectiveness of TENS in the management of pelvic pain related to endometriosis, but they are of uneven quality.
* Evaluating the effectiveness of TENS in the management of endometriosis-related pain under the best methodological conditions remains essential.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 18 years
2. Endometriosis and/or adenomyosis diagnosed by imaging and/or histology
3. Undergoing continuous, stable, and functional hormone treatment (with no menstruation) for at least 2 months
4. No change in hormone treatment planned for the duration of the study
5. Chronic pelvic pain for more than 6 months
6. Pelvic pain at least equal to 2 out of 3 (on the intensity scale: "0 - None," "1 - Mild," "2 - Moderate," "3 - Severe")
7. Agreeing to participate in the study
8. Agrees to limit pain relief treatment during the study to level I painkillers paracetamol and Acupan® (nefopam), and the NSAID Antadys® (flurbiprofen)
9. Has a computer, tablet, or cell phone with an internet connection
10. Is affiliated with a social security system or is a beneficiary of such a system

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Menopausal women
3. Patients who, in the investigator's opinion, have experienced an acute worsening of endometriosis symptoms in the last 28 days
4. Patients with altered sensitivity in the area where the device is applied (hypoesthesia)
5. Skin allergy to the gel or electrodes
6. Dermatological problem in the stimulation area
7. Patients with an implanted pacemaker or active implanted medical device.
8. Epilepsy
9. Current thrombophlebitis or arterial thrombosis
10. Cancer or malignant disease with an expected survival of < 12 months
11. Alcoholism or drug addiction
12. Fibromyalgia
13. Women who have already tried TENS
14. Patients unable to understand and use the English language to communicate fluently
15. Patients with cognitive impairments
16. Untreated severe psychiatric illness and/or psychological condition that is the primary determinant of the patient's condition
17. Participation in another intervention study that may impact the results of the current study
18. Patient using > 90 morphine equivalents/day (at least once in the last 28 days)
19. Gynecological and/or endometriosis surgery planned within the next 3 months
20. History of endometriosis surgery within the last 6 months
21. Patient who has undergone a hysterectomy or bilateral oophorectomy
22. Patient under legal protection (guardianship or conservatorship) or patient deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the mean value of average pain | 56 days
  Change in the mean value of average pain over the previous 24 hours, measured daily during the P1 investigation phase (between D1 and D28±2), compared with the run-in period (between D-35 and D-8).
  Participants will assess their average pain over the past 24 hours on a 100 mm visual analog scale (VAS) every day. The average of these daily values will be calculated over the run-in period (between D-35 and D-8), during the P1 investigation phase (between D1 and D28±2), and during the P2 extension phase (between D29±2 and D56±2). The visual analog scale will be available on the data collection tool/website provided and accessible throu PC, tablet or smartphone. The VAS is presented as a 100 mm horizontal line with no boundaries, marked at the left end with "no pain" and at the other end with "worst pain imaginable." Repeated pain measurements during the run-in period will provide a reliable baseline value that takes into account daily variations.

CONTACTS AND LOCATIONS:
Overall Officials: Bejamin MERLOT, Principal Investigator — IFEM Endo, Clinique Tivoli-Ducos, 5 rue Auguste Poirson, 33000 Bordeaux, France
Locations (1):
- IFEM Endo, Clinique Tivoli-Ducos, Bordeaux, France